CLINICAL TRIAL: NCT00099983
Title: CSP #504 - Risperidone Treatment for Military Service Related Chronic Post-Traumatic Stress Disorder
Brief Title: Risperidone Treatment for Military Service Related Chronic Post Traumatic Stress Disorder
Acronym: CSP #504
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 504
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Stress Disorders; Post-Traumatic
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone (Active Comparator): 1 mg/day tablet for week one, increasing by 1 mg/day weekly to a target dose of 3 mg/day to a maximum of 4 mg/day allowed after a minimum of 4 weeks at the target dose 3 mg/day
  Interventions: Drug: Risperidone
- Sugar Pill (Placebo Comparator): Placebo 1 mg/day tablet for week one, increasing by 1 mg/day weekly to a target dose of 3 mg/day to a maximum of 4 mg/day allowed after a minimum of 4 weeks at the target dose 3 mg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — Initiate treatment with a low dose (1 mg/day HS) for week one, increasing by 1 mg/day weekly to a target dose of 3 mg/day. Escalation to a maximum of 4 mg/day will be allowed after a minimum of 4 weeks at the target dose (3 mg/day). Reduction to a lower dose will be allowed at any time, based on adverse effects. Treatment will continue for 6 months. Patients who discontinue treatment will be allowed to resume treatment at any time.
  Other Names: Risperdal
  Arms: Risperidone
Drug: Placebo — Placebo
  Other Names: Suger Pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this research of 400 participants is to determine whether a drug called risperidone can decrease symptoms of Post-Traumatic Stress Disorder (PTSD). It is a placebo-controlled study, meaning that half of the participants will be assigned to receive a pill that contains no drug. The treatment phase of the study will last for 6 months, during which time participants will continue to receive all their usual treatments in addition to the study treatment and will be asked to complete procedures and assessments (questionnaires, interviews, laboratory tests, physical exams, etc.) related to their PTSD symptoms at various points within the 6-month treatment phase. At the end of the 6-month study, participants will discontinue the study treatment.

DETAILED DESCRIPTION:
Primary Hypothesis: Risperidone will reduce symptoms of PTSD, relative to placebo, in veterans with military service related chronic PTSD who have been partial or non-responders to antidepressant medications.

Secondary Hypothesis: Risperidone is safe and well-tolerated in veterans with military service related chronic PTSD, and patients will comply with its prescription. As a result, patients will show improvement in the secondary consequences of PTSD for the veteran and for the VA.

Intervention: Usual (PTSD) care plus Risperidone vs usual (PTSD) care plus placebo Study Abstract: Four hundred veterans with the diagnosis of military-related PTSD will be enrolled at 20 VAMC hospitals over a two-year period. An equipoise stratification design will be used to randomize patients in a double-blind manner to risperidone or placebo (~200 patients in each group) for six months of treatment. Usual care will be provided for all patients for treatment of PTSD and other psychiatric and medical disorders. Comparisons between the risperidone and placebo groups will be made at the end of six months to answer the primary question. The sample size is calculated to give 90% power at the two-sided alpha level of 0.05 for the overall test for the CAPS score change.

STUDY UPDATE/NOTES: The study kicked-off in late July 2006 with recruitment expected to begin October 1, 2006.

Oct2006 - Participating sites are seeking approval for the protocol amendment which resulted from the Kick-Off meeting. Patient recruitment at each site will begin as soon as they receive approval of the amendment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Military service related chronic PTSD
* CAPS score >50
* Participant in VA outpatient PTSD clinic
* History of non-response to two or more antidepressants

Exclusion Criteria:

* Comorbid Axis I diagnosis requiring antipsychotic medication
* Substance dependence diagnosis (excluding nicotine)
* Hepatic or renal problems
* Incompatible medical diagnosis or medication (i.e., coumadin, insulin)
* Unstable living arrangements
* Assault or suicide gesture within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Krystal, Study Chair — VA Connecticut Health Care System (West Haven)
Locations (20):
- United States (20):
  - VA Medical Center, Tuscaloosa, Tuscaloosa, Alabama
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, Miami, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Providence, Providence, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - Central Texas Veterans Health Care System, Temple, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Krystal JH, Pietrzak RH, Rosenheck RA, Cramer JA, Vessicchio J, Jones KM, Huang GD, Vertrees JE, Collins J, Krystal AD; Veterans Affairs Cooperative Study #504 Group. Sleep disturbance in chronic military-related PTSD: clinical impact and response to adjunctive risperidone in the Veterans Affairs cooperative study #504. J Clin Psychiatry. 2016 Apr;77(4):483-91. doi: 10.4088/JCP.14m09585. PMID 26890894
- [Derived] Krystal JH, Rosenheck RA, Cramer JA, Vessicchio JC, Jones KM, Vertrees JE, Horney RA, Huang GD, Stock C; Veterans Affairs Cooperative Study No. 504 Group. Adjunctive risperidone treatment for antidepressant-resistant symptoms of chronic military service-related PTSD: a randomized trial. JAMA. 2011 Aug 3;306(5):493-502. doi: 10.1001/jama.2011.1080. PMID 21813427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited initially from 20 VA Medical Centers over a 2-year period. To address low recruitment rates and other issues, 8 sites were discontinued and 6 sites were added during the course of the study.
Groups:
- Risperidone: an atypical antipsychotic indicated for the treatment of schizophrenia but not for Post Traumatic Stress Disorder (PTSD). Some of additional unlabeled uses of risperidone include behavioral symptoms associated with dementia in the elderly, bipolar disorder, Tourette's disorder, pervasive developmental disorder and autism.
  (1 mg/day HS) for week one, increasing by 1 mg/day weekly to a target dose of 3 mg/day. Escalation to a maximum of 4 mg/day will be allowed after a minimum of 4 weeks at the target dose (3 mg/day).
- Sugar Pill: Placebo Sugar Pill 1 mg/day HS) for week one, increasing by 1 mg/day weekly to a target dose of 3 mg/day. Escalation to a maximum of 4 mg/day will be allowed after a minimum of 4 weeks at the target dose (3 mg/day).
Period: Overall Study
Arm/Group | Risperidone | Sugar Pill
Started | 147 | 149
Completed | 123 | 124
Not Completed | 24 | 25
Not completed — Lost to Follow-up | 2 | 3
Not completed — Missing Source Documents | 14 | 15
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Unable to return for appointments | 1 | 1
Not completed — Moved | 1 | 0
Not completed — Other psychiatric problem | 1 | 0
Not completed — Incarcerated | 0 | 1
Not completed — Intolerant of burden of visits | 0 | 1
Not completed — Other issue | 1 | 0

BASELINE CHARACTERISTICS:
Population: Valid diagnostic baseline data were collected on 267 patients randomized to receive risperidone (n=133) and placebo (n=134). The 29 patients with "missing source documents" as reported in Participant Flow were not included in any analyses.
Groups:
- Risperidone: Risperidone : atypical antipsychotic
- Sugar Pill: PTSD
  Placebo : Placebo
- Total: Total of all reporting groups
Arm/Group | Risperidone | Sugar Pill | Total
Number analyzed (Participants) | 133 | 134 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 134 | 267
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.8) | 54.5 (10.6) | 54.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 128 | 130 | 258
Region of Enrollment [Number; unit: participants]
  United States | 133 | 134 | 267

OUTCOME MEASURES:

1. Primary Outcome: Change in CAPS Score From Baseline to Week 24
Description: The primary outcome measure for this study was the total score on the 34-item Clinician-Administered PTSD Scale (CAPS). This study was the intent-to-treat analysis of the improvement in PTSD symptoms from baseline to week-24 follow-up as measured by the CAPS. Total score range for the CAPS is 0-136 with higher values representing a worse outcome. This study was powered initially to detect a 9-point difference between the treatment groups in the CAPS change score.
Time Frame: 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risperidone | Sugar Pill
Number analyzed (Participants) | 123 | 124
units on a scale | -16.3 [-19.7 to -12.9] | -12.5 [-15.7 to -9.4]

ADVERSE EVENTS:
Time Frame: Within 72 hours of site being made aware of event.
Arm/Group | Risperidone | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 16/133 | 10/134
Other Adverse Events (participants affected / at risk) | 0/133 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone (N=133) | Sugar Pill (N=134)
Suicidal ideation (Psychiatric disorders) | 8 (8) | 2 (2)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Gastrooesphageal reflus Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Infections (Infections and infestations) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes